CLINICAL TRIAL: NCT06513416
Title: Gut Microbiota and Pulmonary Complications After Non Cardiac Elective Surgery in Elderly Patients
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Huang YuGuang, Chief physician, Peking Union Medical College Hospital
Other Study IDs: K5484
Record Dates: First submitted 2024-07-17; First posted 2024-07-22 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Gut Microbiota; Postoperative Pulmonary Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PPCs+ group: Patients who experienced postoperative pulmonary complications belong to the PPC positive group
  Interventions: Procedure: Elective upper abdominal surgery
- PPCs- group: Patients who experienced no postoperative pulmonary complications belong to the PPC negative group
  Interventions: Procedure: Elective upper abdominal surgery

INTERVENTIONS:
Procedure: Elective upper abdominal surgery — The included elderly patients are those who are preparing for elective upper abdominal surgery and the surgery time exceeds 2 hours.

SUMMARY:
This study adopts a combination of retrospective and prospective cohort research methods to explore the composition of preoperative oropharyngeal and gut microbiota in elderly patients undergoing elective upper abdominal surgery, aiming to analyze the correlation between preoperative oropharyngeal and intestinal microbiota composition and metabolite levels and the occurrence of postoperative pulmonary complications (PPCs). The research subjects of the retrospective cohort study were participants (ClinicalTrials.gov No. NCT05679661) included in the prospective RCT on the effects of perioperative immune nutrition intervention and oral hygiene on postoperative complications in elderly patients, which was conducted at Peking Union Medical College Hospital from January 2023 to present. The prospective cohort study plans to continue enrolling elderly patients aged ≥ 65 who underwent elective upper abdominal surgery.

This study collects preoperative oropharyngeal and fecal samples, as well as preoperative plasma from patients for microbial sequencing and untargeted metabolomics analysis. The main outcome measurement is PPCs, which include pneumonia, atelectasis, and hypoxemia within 7 days after surgery. Inflammatory cells and cytokines in peripheral blood are secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 65 years old;
2. Surgery: Upper abdominal surgery (expected duration ≥ 2 hours);
3. Anesthesia methods: general anesthesia, tracheal intubation;
4. ASA classification: I-IV levels;
5. Postoperative Pulmonary Complications Risk Score (ARISCAT): Medium to High Risk
6. Patients or their families are able to understand the research protocol and are willing to participate in this study, providing written informed consent

Exclusion Criteria:

1. Emergency surgery;
2. This is the second surgery within the past month;
3. Preoperative presence of pulmonary infection or other serious pulmonary complications
4. Patients who have used antibiotics, probiotics, and acid suppressants within one month before surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients over 65 years old who plan to undergo elective upper abdominal surgery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with postoperative pulmonary complications | Within 7 days after surgery
  Including pneumonia, atelectasis, and hypoxemia

SECONDARY OUTCOMES:
Number of inflammatory cells in peripheral blood before and after surgery | Before and within 7 days after surgery
  Inflammatory cells include white blood cells, neutrophil count, and lymphocyte count
Concentration of inflammatory cytokines in peripheral blood before and after surgery | Before and within 7 days after surgery
  Inflammatory factors include high-sensitivity C-reactive protein (CRP) and procalcitonin (PCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided